CLINICAL TRIAL: NCT04795687
Title: Association of Metagenomics and Transcriptomics With the Appearance and Evolution of an Ischemic Stroke
Brief Title: Discovering Patterns in the Gut Microbiota Associated With the Risk of Stroke and the Outcome After a Stroke and Integration of These Data With Genomic Information to Find New Drug Targets and New Treatments to Improve Neurological Evolution and Functional Status of Stroke Patients.
Acronym: MAESTRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: IIBSP-MAE-2020-12
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Stroke
Keywords: Gut microbiota; Stroke; Metagenomics
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and fecal samples stored with ethanol 96%.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemic stroke patients
- Control

SUMMARY:
The composition of the intestinal microbiota is associated with the risk of stroke and with post-stroke neurological evolution. At the same time, the genetics and epigenetics of each patient are associated with the composition of the intestinal microbiota. The study of the microbiome in stroke patients will allow finding new therapeutic targets for the treatment of stroke patients.

For the study, samples will be collected from those patients with ischemic stroke who come to the hospital while the study is being carried out, taking into account certain criteria: the patients must be over 18 years of age, have suffered an ischemic stroke (demonstrated by resonance or head CT), not have any additional serious illness or unstable medical condition, and not be included in clinical trials with neuroprotective drugs. On the other hand, the control group will be asymptomatic, and will be made up of people who have not previously suffered a stroke or a cardiovascular event and who do not have diseases that affect the digestive tract.

The main variables of the study are the risk of stroke and disability after a cerebrovascular accident (measured by mRS at 3rd month). Microbiota, genetic and epigenetic variables are also taken into account, such as the presence and levels of bacteria, dysbiosis, genetic polymorphisms and levels of methylation in CpG islands.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke (demonstrated by resonance or head CT).

Exclusion Criteria:

* Patients under 18 years of age.
* Additional serious illness or unstable medical condition.
* Inclusion in clinical trials with neuroprotective drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples will be collected from those patients with ischemic stroke who attend the Hospital de la Santa Creu i Sant Pau while the study is carried out.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of stroke and disability after a stroke | 3 months
  Use of the Modified Rankin Scale (mRS), evaluted from 0 to 6 (where higher scores mean worse outcome), to asses disability in patients who have suffered a stroke and comparison over time to check for recovery and degree of continued disability

CONTACTS AND LOCATIONS:
Overall Officials: Israel Fernández Cadenas, PhD, Principal Investigator — Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Institut de Recerca Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD).
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: IPD will be shared for further analysis under request. Requests will be reviewed by the overall study official Dr. Israel Fernández Cadenas.

REFERENCES:
- [Derived] Lledos M, Prats-Sanchez L, Muino E, Cullell N, Llucia-Carol L, Carcel-Marquez J, Gallego-Fabrega C, Martin-Campos JM, Marin R, Aguilera-Simon A, Guasch-Jimenez M, Ezcurra-Diaz G, Camps-Renom P, Del Mar Freijo M, Marti-Fabregas J, Fernandez-Cadenas I. Influence of the Gut Microbiota on Acute Ischemic Stroke Functional Outcomes at Three Months. Eur J Neurol. 2025 Jul;32(7):e70265. doi: 10.1111/ene.70265. PMID 40686474